CLINICAL TRIAL: NCT01955564
Title: A Phase I, Prospective, Randomized, Double-blind, Placebo-controlled, Sequential-cohort, Escalating, Single-dose Study Designed to Determine the Maximum Tolerated Oral Dose of NW-3509A in Healthy, Male Volunteers.
Brief Title: A Phase I- Sequential Cohort Dosing to Determine Maximum Tolerated Dose in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NW-3509A/001/I/2011
Record Dates: First submitted 2013-08-21; First posted 2013-10-07 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1 (Experimental): NW-3509a - 1mg or placebo
  Interventions: Drug: NW-3509a
- Cohort 2 (Experimental): NW-3509a 2mg or placebo
  Interventions: Drug: NW-3509a
- Cohort 3 (Experimental): NW-3509a 5mg or placebo
  Interventions: Drug: NW-3509a
- Cohort 4 (Experimental): NW-3509a 10 mg or placebo
  Interventions: Drug: NW-3509a
- Cohort 5 (Experimental): NW-3509a 20 mg or placebo
  Interventions: Drug: NW-3509a
- Cohort 6 (Experimental): NW-3509a 30 mg or placebo
  Interventions: Drug: NW-3509a

INTERVENTIONS:
Drug: NW-3509a — single dose
  Other Names: NW-3509

SUMMARY:
This is a prospective, 8-day, randomized, double-blind, placebo-controlled, sequential-cohort study designed to evaluate the safety, tolerability, and MTD of single escalating oral doses of NW-3509A in healthy male volunteers. Six independent cohorts of 12 volunteers each will participate in this study, with the first 9 volunteers in each cohort to qualify being randomized to receive study medication and the remaining 3 to be used as backups/ alternates. In each cohort, 6 subjects will be randomly assigned to receive NW-3509A and 3 subjects will receive placebo.

DETAILED DESCRIPTION:
Doses from 1 to 30 mg were tested

ELIGIBILITY:
Inclusion Criteria:

* Demographics

Volunteers will meet the following demographic inclusion criteria:

1. Age - between 18 and 45 years of age, inclusive.
2. Sex - males.
3. The subject has a body weight of at least 45 kg and a body mass index of ≤30.

   Procedural

   Volunteers will meet the following procedural criteria:
4. They are cooperative, able to take oral medication, willing to complete all aspects of the study, and capable of doing so.
5. They will be able to understand the instructions and fully participate.
6. They will have provided written informed consent prior to participating in the study.
7. The subject is in good health with no history of significant medical disease as determined by the investigator.

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment:

General Medical Status

1. An advanced, severe, or unstable disease of any type that may interfere with any of the study evaluations, including any medical condition that could be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical or mental status of the volunteer to a significant degree or put the volunteer at special risk (e.g., liver or kidney disease; malignancy);
2. A disability that may prevent the volunteer from completing all study requirements (e.g., blindness, deafness, severe language difficulty);
3. A current diagnosis of active, uncontrolled peptic ulceration within the last year;
4. A current diagnosis of acute, severe, or unstable asthmatic condition.

   Cardiovascular
5. A current diagnosis of severe or unstable cardiovascular disease;
6. A current diagnosis of sick-sinus syndrome or conduction deficits (e.g., sino-atrial block (<0.22), second or third degree atrio-ventricular block);
7. Any history or current evidence of a cardiac illness as determined by the investigator;
8. Any clinically significant ECG abnormality, including a disorder of rate, rhythm, or conduction, or other morphological changes, or a QTcF interval (Fridericia's correction formula) on the ECG >450 msec. The 12-lead ECG will be used for determining the suitability of the subject for inclusion in the study (determined by the investigator);
9. Vital signs (supine) outside the following ranges:

   * Systolic blood pressure below 100 or above 139 mmHg;
   * Diastolic blood pressure below 50 or above 89 mmHg;
   * Radial pulse below 50 or above 90 bpm.

   CNS related
10. Any history or current diagnosis of any neurodegenerative illness;
11. History or current diagnosis of epilepsy or seizure disorder.

    Psychiatric
12. Any past or current psychiatric illness (DSM-IV-TR Axis 1 diagnosis);
13. Subjects with current or past suicidal ideation.

    Study-specific criteria
14. History of serious adverse reactions or hypersensitivity to any drug;
15. Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis);
16. Alcohol or drug abuser; currently or at any time in the last 5 years;
17. Abnormal physical findings of clinical significance at the screening examination or baseline that would interfere with the objectives of the study;
18. Need of any prescription medication within 14 days prior to the administration of the study drug, and/or non-prescription medication within 7 days prior to the administration of the drug;
19. Participation in other clinical trials during the last 2 months in which an investigational drug or a commercially available drug was tested;
20. Loss of 500 ml or more of blood during the 3-month period before the study, e.g. as a donor.
21. Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, inflammatory bowel disease, chronic symptoms of pronounced constipation or diarrhea, or conditions associated with total or partial obstruction of the urinary tract;
22. Symptoms of a significant somatic or mental illness in the four-week period preceding study drug administration;
23. History of hepatitis B and/or C, and/or positive serology results, which indicate the presence of hepatitis B and/or C (Hepatitis B surface antigen and/or antibody to Hepatitis C);
24. Positive results from the HIV serology;
25. Positive results of the drug and alcohol tests at screening and/or check-in at the unit;
26. Smoker; currently or at any time in the last 5 years;

    Laboratory abnormalities
27. Clinically significant abnormalities in routine laboratory examinations (hematology; blood chemistry, including electrolytes and liver and kidney function tests; urinalysis), as determined by the Principal Investigator in consultation with the Sponsor, at the screening evaluation;
28. Clinically important laboratory abnormalities in thyroid function tests at screening:

    • TSH > 8.0 mU/L and/or Free T4 < 9 pmol/L;

    Concomitant therapy
29. A known exaggerated pharmacological sensitivity or hypersensitivity to drugs similar to NW-3509A. Possible examples are volunteers who have experienced hypersensitivity reactions to sodium channel blockers;
30. Ingested any of the following substances:

    * An investigational drug during the past 2 months;
    * A drug or treatment known to cause major organ system toxicity during the past year;
    * Any prescription drug or OTC product if taken continuously (Medical Monitor from Newron should be contacted if the Investigator wants to include a volunteer who is taking an OTC product);
    * Alcohol intake should be limited to 2 drinks per day during the 2 weeks prior to dosing; alcohol consumption will be prohibited from 72 hours prior to admittance on Day -1 through to the final safety evaluations on Day 8.
    * Caffeine-containing products should be limited (equivalent of 2 cups of coffee per day) during the 2 weeks prior to dosing and through to the final safety evaluations on Day 8.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Leibowitz, MD, Principal Investigator — Collaborative Neuroscience Network Phase I Unit; Ravi Anand, MD, Study Director — Newron Pharmaceuticals SPA
Locations (1):
- Collaborative Neuroscience Network-Clinical Pharmacology Unit, Long Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 54 healthy males, who were between the age of 18-45 years old, with a minimum body weight of 45 kg and body mass index of more than or equal to 30, were recruited and observed in the period from 23rd of July 2013 till 19th of September 2014 in this study conducted at a single site in the US.
Groups:
- Placebo: Placebo, single dose
- Cohort 1: NW-3509a - 1mg, single dose
- Cohort 2: NW-3509a 2mg, single dose
- Cohort 3: NW-3509a 5mg, single dose
- Cohort 4: NW-3509a 10 mg, single dose
- Cohort 5: NW-3509a 20 mg, single dose
- Cohort 6: NW-3509a 30 mg, single dose
Period: Overall Study
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 18 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 18 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 9 healthy volunteers were assigned per cohort, within which 6 subjects received NW-3509A and 3 subjects received placebo by randomised selection.
Groups:
- Placebo: placebo: single dose
- Cohort 1: NW-3509a - 1mg
  NW-3509a: single dose
- Cohort 2: NW-3509a 2mg
  NW-3509a: single dose
- Cohort 3: NW-3509a 5mg
  NW-3509a: single dose
- Cohort 4: NW-3509a 10 mg
  NW-3509a: single dose
- Cohort 5: NW-3509a 20 mg
  NW-3509a: single dose
- Cohort 6: NW-3509a 30 mg NW-3509a: single dose
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Total
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 54
Age, Customized [Mean (Standard Deviation); unit: years]
  18-45 | 31.27 (7.71) | 28.33 (6.31) | 23.83 (6.91) | 30.33 (8.12) | 34.83 (5.85) | 29.50 (3.51) | 24.33 (3.56) | 28.92 (3.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 54
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 0 | 1 | 1 | 2 | 2 | 0 | 8
  African American | 7 | 2 | 4 | 4 | 3 | 4 | 1 | 25
  Asian | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 5
  Caucasian | 8 | 2 | 1 | 1 | 0 | 0 | 3 | 15
  Native American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 54

OUTCOME MEASURES:

1. Primary Outcome: Physical Examination Shift Table
Description: Physical examinations were carried out on the following: Lymph nodes, mouth, neck, nervous system, nose, skin and throat.
Time Frame: Day -1(pre-dose) through Day 8 (Discharge)
Measure: Number; unit: Participants abnormal at end of study
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6
Participants abnormal at end of study | 1 | 1 | 0 | 0 | 1 | 1 | 0

2. Secondary Outcome: Maximum Plasma Concentration of NW-3509A at Doses Tested
Description: Plasma concentration data, derived PK parameters, and urine data are summarized as maximum plasma concentration (Cmax).
  The plasma concentrations of NW-3509A in the samples taken from the subjects receiving placebo were below the limit of quantification (<1.00 ng/mL) in all cases (n=18).
Time Frame: Baseline up to 32 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 1: NW-3509a 1mg, single dose
- Cohort 4: NW-3509a 10mg, single dose
- Cohort 5: NW-3509a 20mg, single dose
- Cohort 6: NW-3509a 30mg, single dose
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 2.08 (1.20) | 3.49 (1.98) | 14.2 (7.2) | 22.5 (16.4) | 36.4 (30.1) | 93.3 (18.0)

3. Secondary Outcome: Total Drug Exposure Over Time (AUC0-t) of NW-3509A at Doses Tested
Description: Plasma concentration data, derived PK parameters, and urine data were summarized as total drug exposure over time (AUC0-t).
  The plasma concentrations of NW-3509A in the samples taken from the subjects receiving placebo were below the limit of quantification (<1.00 ng/mL) in all cases (n=18).
Time Frame: Baseline up to 32 hours post-dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng.h/mL | 6.71 (9.24) | 13.4 (11.2) | 56.7 (30.5) | 101 (86) | 166 (175) | 350 (34)

ADVERSE EVENTS:
Time Frame: Adverse Event evaluations were performed during the screening period, at baseline, Day 2 and Day 8. In addition, all subjects were followed up for 30 days after their dose of study medication for the occurrence of any SAEs
Description: Systematic assessment by standard questionnaires, regular investigator assessment, and regular laboratory testing at each visit.
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/18 | 3/6 | 1/6 | 3/6 | 2/6 | 5/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Cohort 1 (N=6) | Cohort 2 (N=6) | Cohort 3 (N=6) | Cohort 4 (N=6) | Cohort 5 (N=6) | Cohort 6 (N=6)
Postural Orthostatic and tachycardia syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — mild
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — mild
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — mild
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — mild
Confusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — mild
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — mild
Excoriation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — mild
Thermal burn (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — mild
Blood creatine phosphate kinase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — mild
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — mild
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — mild
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — mild
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — mild
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — mild and moderate
Presyncope (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — mild
Somnolence (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — mild and moderate
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — mild and moderate
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — mild
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — mild
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No